CLINICAL TRIAL: NCT03724903
Title: Ductal Lavage Versus Corticosteroids Therapy for Idiopathic Granulomatous Mastitis: a Multicenter, Randomized, Open-labelled, Non-inferior Trial.
Brief Title: Ductal Lavage Versus Corticosteroids Therapy for Idiopathic Granulomatous Mastitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chen Kai, Dr., Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ductal-2018-Jun-14
Record Dates: First submitted 2018-10-28; First posted 2018-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-01

CONDITIONS: Granulomatous Mastitis
MeSH Terms: conditions — Granulomatous Mastitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ductal lavage (Experimental): Ductal lavage and breast massage for two weeks.
  Interventions: Procedure: Ductal lavage
- Corticosteroids therapy (Active Comparator): Oral corticosteroids therapy for 6 months.
  Interventions: Drug: Corticosteroid therapy

INTERVENTIONS:
Procedure: Ductal lavage — The patients received ductal lavage and breast massage every other day for two weeks. We used lidocaine (1%) for local anesthesia around the nipple. We used a lacrimal probe to identify 4-5 openings in the lactiferous ducts on the nipple and inserted the infusion cannula (21-23G). A total of 25ml of irrigation solution (5 ml of 2% lidocaine, 40 mg of triamcinolone acetonide, 20 ml of 0.9% saline and 1.0 g of ceftriaxone) was pumped into the ducts over 20-25 minutes. The patient returned to the clinic the next day for breast massage, and the cycle was repeated for two weeks.
  Arms: Ductal lavage
Drug: Corticosteroid therapy — Methylprednisolone(Common brand names: Medrol) or prednisone 20-40mg, qd for two weeks, then temper the dose gradually, and then 20mg qd for maintenance (The total duration of the treatment is 6 months).
  Arms: Corticosteroids therapy

SUMMARY:
A single-arm, proof-of-concept trial has shown the safety and efficacy of ductal lavage as a treatment for idiopathic granulomatous mastitis patients (Manuscript accepted in Journal of Surgical Research 2018). In this multicenter, randomized, open-labeled, non-inferior trial, the investigators are going to enroll eligible granulomatous mastitis patients and randomized them into ductal lavage versus. corticosteroids therapy group. The primary endpoint of this study is the complete clinical response rate at 1 year after the enrollment. The aim of this study is to provide evidence for the management of idiopathic granulomatous mastitis patients .

DETAILED DESCRIPTION:
Non-lactational mastitis (NLM) consists of a broad spectrum of inflammatory breast diseases. Among them, periductal mastitis and idiopathic granulomatous mastitis(IGM) are the most commonly encountered in clinical practice. IGM can be diagnosed when all possible causes of granulomatous diseases (known mycobacterial or fungal infection, Wegener granulomatosis, sarcoidosis, etc.) are excluded. There is no consensus on the standard treatment of IGM patients. Surgery, oral corticosteroids, topical steroids, immunosuppressive therapy, and observation alone were all proposed as the treatment for IGM patients. However, all of the evidences are derived from retrospective studies. In a previous study, the investigators conducted a single-arm, proof-of-concept trial that showed the safety and efficacy of ductal lavage as a treatment for IGM patients. Ductal lavage is possible to spare the patients from corticosteroids therapy and or surgery. To further address this issue, the investigators are going to conduct this multicenter, randomized, open-labeled, non-inferior trial, to compare the efficacy and safety of ductal lavage and corticosteroids therapy. The aim of this study is to provide evidence for the management of IGM patients.

ELIGIBILITY:
Inclusion Criteria:

* Female, age between 18 and 65 years old.
* Inform consent signed.
* Clinical diagnosis of non-lactating mastitis, defined as mastitis occurred more than 1 month after the cessation of lactation.
* Clinical and pathological diagnosis of idiopathic granulomatous mastitis.
* Never receive surgical treatments, or corticosteroids therapy after the cessation of lactation. Core needle biopsy is allowed.
* Good health, judged by clinicians, to receive ductal lavage.
* M score >=2

Exclusion Criteria:

* Grade III inverted nipple(Plastic. Reconstruction. Surgery. 104: 389, 1999.)
* Lactational mastitis patients.
* Bilateral IGM patients.
* Clinically diagnosis of periductal mastitis.
* Pathological diagnosis of breast carcinoma.
* Pregnant women.
* Evidences suggest possible diagnosis of SLE(systemic lupus erythematosus), rheumatic disorders or other systematic auto-immune diseases.
* Evidences suggest possible diagnosis of tuberculosis.
* Evidences suggest possible diagnosis of fungus infection of the breast
* History of breast trauma.
* History of taking oral corticosteroids or anti-tuberculosis treatment.
* Imaging examinations indicates foreign objects retained in the breast
* Presence of sepsis or severe inflammation caused by IGM, for which surgery is likely required.
* Patients with inappropriate coagulation function, cardiac function, pulmonary function, liver and renal function, that clinicians judges as not suitable to participate in this study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Complete Clinical Response(cCR) | 1 year since randomization
  The proportion of patients that achieve M-score <=1 at 1 year after the treatment.

SECONDARY OUTCOMES:
Time to cCR | 1 year since randomization
  The median time to cCR since the randomization.
Treatment failure (TF) rate | 1 year since randomization
  The proportion of patients with TF at 1 year since the randomization. The TF status is defined as the following:
  1. If the patient has M-score>=6 before randomization, TF is defined as the M-score still remains >=6 at one month since the randomization.
  2. If the patient has M-score between 4 and 5 before randomization, TF is defined as the M-score still remains at >=4, and never have been lower than 4.
  3. If the patient has M-score<4 before randomization, and never reaches cCR since randomization, and during follow-up, the M-score is found to be >5 and last for one month.
Relapse rate | 1 year since randomization
  The proportion of patients that had M-score>4 among those patients who achieved cCR.
Adverse events | 1 year since randomization
  Pre-defined and any other unexpected adverse events would be recorded and compared between the two arms.
Protocol compliance rate | 1 year since randomization
  The proportion of patients who received the treatment protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Erwei Song, MD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (2):
- China (2):
  - Jiangmen Maternal and Child Health Care Population ＆ Family Planning Service Center, Jiangmen, Guangdong
  - Lian Jiang People'S Hospital, Lianjiang, Guangdong

IPD SHARING:
Plan to Share IPD: No
The study protocol and the raw and clean data for analysis will be shared among the participated researchers. Non-researchers could obtain relevant informations from the researchers upon reasonable requests.

REFERENCES:
- [Background] Hu T, Li S, Huang H, Huang H, Tan L, Chen Y, Deng H, Wu J, Zhu L, Zhang J, Su F, Chen K. Multicentre, randomised, open-label, non-inferiority trial comparing the effectiveness and safety of ductal lavage versus oral corticosteroids for idiopathic granulomatous mastitis: a study protocol. BMJ Open. 2020 Oct 10;10(10):e036643. doi: 10.1136/bmjopen-2019-036643. PMID 33039992
- [Background] Chen K, Zhu L, Hu T, Tan C, Zhang J, Zeng M, Li S, Song E. Ductal Lavage for Patients With Nonlactational Mastitis: A Single-Arm, Proof-of-Concept Trial. J Surg Res. 2019 Mar;235:440-446. doi: 10.1016/j.jss.2018.10.023. Epub 2018 Nov 19. PMID 30691827
- [Derived] Chen X, Huang H, Huang H, Yong J, Zhu L, Chen Q, Tan L, Zeng Y, Yang Y, Zhao J, Rao N, Ding L, Wu W, Li Y, Gui X, Ye L, Xu Y, Jiang Y, Su L, Xiao Q, Cai X, Hu T, Tan C, Liu Q, Liu S, Zhao J, Wang Y, Yu F, Zhang J, Li S, Chen K. Ductal lavage followed by observation versus oral corticosteroids in idiopathic granulomatous mastitis: A randomized trial. Nat Commun. 2024 Oct 23;15(1):9144. doi: 10.1038/s41467-024-53143-2. PMID 39443446